CLINICAL TRIAL: NCT02231970
Title: Endoscopic Sleeve Gastroplasty for Treatment of Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo Hospital de Madrid (Other)
Responsible Party: Principal Investigator, Sofia Perea, Director Clinical Trials Unit., Director, Clinical Trial Unit, Grupo Hospital de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 657-GHM
Record Dates: First submitted 2014-09-01; First posted 2014-09-04 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Obesity
Keywords: Obesity; Endoscopic sleeve gastroplasty; Weight loss
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endoscopic sleeve gastroplasty (Experimental): The intervention is an endoscopic procedure: to perform endoscopic sleeve gastroplasty we used a cap-based flexible endoscopic suturing system (OverStitch™, Apollo, Inc. Austin, Texas) mounted on a double-channel endoscope (GIF-2T160; Olympus Medical Systems Corporation, Tokyo, Japan) to achieve full-thickness, running sutures through the gastric wall from antrum to fundus.
  Interventions: Procedure: Endoscopic sleeve gastroplasty

INTERVENTIONS:
Procedure: Endoscopic sleeve gastroplasty — To perform endoluminal gastric volume reduction by the Endoscopic sleeve gastroplasty
  Other Names: ESG

SUMMARY:
Emerging endoscopic techniques are minimally invasive and can mimic the anatomic alterations achieved by surgical sleeve gastrectomy.

The study hypothesis is if endoscopic sleeve gastroplasty is effective and useful in the treatment of patients with obesity

DETAILED DESCRIPTION:
The endoscopic sleeve gastroplasty method to perform endoluminal gastric reduction were by a cap-based flexible endoscopic suturing system. Post procedure care includes close follow-up by a nutritionist and a psychologist weekly.The outcome assessment included: change in body weight, percentage of loss of excess body weight and adverse effects

ELIGIBILITY:
Inclusion Criteria:

Obesity Willingness and ability of patients to be treated by a multidisciplinary team for at least 1 year -

Exclusion Criteria:

Prior endoscopy discarded patients with gastric findings (potentially bleeding lesions and neoformative findings ) Coagulopathy Psychiatric disorders

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | One year

SECONDARY OUTCOMES:
Safety | One year
  Any complications following the intervention like abdominal pain or bleeding

OTHER OUTCOMES:
Percentage of excess weight loss | One year
  Percentage of excess weight loss defined as the percentage of weight loss in relation with initial weight minus weight at BMI of 25 kg/m2

CONTACTS AND LOCATIONS:
Overall Officials: GONTRAND LOPEZ-NAVA, MD, Principal Investigator — HOSPITAL UNIVERSITARIO SANCHINARRO
Locations (1):
- Hospital Universitario Sanchinarro, Madrid, Madrid, Spain